CLINICAL TRIAL: NCT07016204
Title: A Randomized Controlled Trial Investigating the Effects of Cognitive-Behavioral Therapy on Neurophysiological and Psychological Outcomes in Individuals With Body Dysmorphic Disorder
Brief Title: CBT Effects on Neurophysiological and Psychological Outcomes in Body Dysmorphic Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Collaborators: Uskudar University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Dr, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INUBDD-CBT-2025
Record Dates: First submitted 2025-06-02; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Body Dysmorphic Disorder
Keywords: Cognitive Behavioral Therapy; BDD; Body Image; EEG; Eye-Tracking; GSR
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants with BDD will be randomly assigned to either a 12-week Cognitive-Behavioral Therapy (CBT) group or a waitlist control group. Neurophysiological and psychometric data will be collected at baseline and post-intervention to evaluate treatment effects.
Masking Description: No masking will be applied. Participants and researchers are aware of group assignments due to the structure of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) Group (Experimental): Participants in this arm will receive 12 sessions of manualized Cognitive-Behavioral Therapy (CBT), each lasting 60 minutes, delivered weekly over 12 weeks. The therapy includes psychoeducation, cognitive restructuring, exposure and response prevention (ERP), mindfulness strategies, and attentional retraining related to appearance concerns.
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Waitlist Control Group (No Intervention): Participants in this arm will receive no active intervention during the 12-week study period but will complete the same neurophysiological and psychometric assessments as the CBT group. After the final follow-up, they will be offered the CBT intervention if desired.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — A structured 12-week psychotherapy protocol targeting maladaptive appearance-related beliefs and behaviors in individuals with Body Dysmorphic Disorder (BDD). The intervention involves individual sessions once per week (60 minutes) and incorporates techniques such as psychoeducation, cognitive restructuring, exposure and response prevention (ERP), mindfulness, and attentional retraining.
  Arms: Cognitive-Behavioral Therapy (CBT) Group

SUMMARY:
This clinical trial aims to investigate how a specific type of psychotherapy called Cognitive-Behavioral Therapy (CBT) can help people who experience Body Dysmorphic Disorder (BDD). BDD is a mental health condition where individuals become excessively preoccupied with perceived flaws in their physical appearance-flaws that are often unnoticeable to others. This distress can interfere significantly with their social, emotional, and daily functioning.

The purpose of this study is to evaluate whether a 12-week CBT program can reduce symptoms of BDD and bring about measurable changes in brain activity, physiological stress responses, and patterns of visual attention when individuals view their own faces or appearance-related images. The researchers will use brainwave recordings (EEG), skin response sensors (GSR), and eye-tracking technology to assess these changes. In addition, participants will complete a set of questionnaires that measure depression, anxiety, emotion regulation, self-esteem, body image beliefs, and self-compassion.

Sixty individuals will take part in the study. Thirty will receive CBT sessions once a week for 12 weeks, while the other thirty will be placed on a waitlist and offered treatment later. The study will compare how symptoms and neurophysiological responses change before and after therapy, and whether these changes differ between those who received immediate treatment and those who did not.

The researchers hypothesize that CBT will reduce emotional distress, improve emotion regulation, and shift brain and body responses toward healthier patterns. This study will help identify how and why therapy works for BDD, and whether technologies like EEG and eye-tracking can be used to monitor treatment progress.

DETAILED DESCRIPTION:
Detailed Description Background and Rationale Body Dysmorphic Disorder (BDD) is a chronic and often severely impairing psychiatric disorder characterized by intrusive preoccupations with perceived flaws in one's appearance-flaws that are often imperceptible to others. Individuals with BDD engage in compulsive behaviors such as mirror checking, grooming, or social avoidance, leading to functional impairment and heightened psychological distress. The condition has a high comorbidity with depression and anxiety, and individuals with BDD are at increased risk for suicidality.

Cognitive-Behavioral Therapy (CBT) is the most evidence-based intervention for BDD, targeting cognitive distortions, avoidance behaviors, and emotional dysregulation related to body image. However, despite robust clinical outcomes, the underlying neurophysiological mechanisms of CBT's effectiveness remain insufficiently explored. This trial seeks to address that gap by integrating behavioral symptom change with objective neurophysiological and attentional measures.

This study investigates whether a structured 12-week CBT program produces measurable improvements in brain function, autonomic nervous system response, and attentional bias among individuals with BDD. By combining EEG, GSR, and eye-tracking methods with validated clinical instruments, the research aims to clarify how therapy modulates both the subjective experience and biological correlates of body image disturbance.

Study Design This is a randomized controlled trial with a pre-post design involving two groups: a CBT intervention group and a waitlist control group. Sixty participants aged 18-50 will be recruited. Thirty participants will meet DSM-5 criteria for BDD and will be randomly assigned to either the CBT intervention group (n=15) or the waitlist control group (n=15). An additional healthy control group (n=30) will serve as a normative baseline for neurophysiological comparisons but will not receive any intervention.

The intervention consists of twelve 60-minute weekly CBT sessions focused on psychoeducation, cognitive restructuring, exposure and response prevention (ERP), mindfulness-based emotional regulation techniques, and attentional retraining exercises.

Experimental Protocol

Participants will undergo pre- and post-treatment assessments that include the following:

Neurophysiological Assessment:

EEG recordings will measure event-related potentials (ERPs) such as N170, P300, Late Positive Potential (LPP), and frontal alpha asymmetry.

GSR will capture sympathetic arousal and recovery rates during exposure to appearance-related stimuli.

Eye-tracking will measure fixation duration, pupil dilation, and gaze patterns toward self-perceived flaws and control features.

Stimuli:

Participants will be exposed to images of their own faces (unaltered, neutral, and digitally altered), appearance-related emotional stimuli (e.g., idealized or distorted faces), and non-threatening neutral or positive stimuli.

After each stimulus, they will rate their distress on a Visual Analog Scale (VAS) ranging from 0 to 10.

Psychometric Assessment:

The following validated self-report and clinician-rated scales will be administered at baseline and post-treatment:

Yale-Brown Obsessive-Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS): Measures the severity of appearance-related obsessions and compulsions.

Body Image Disturbance Questionnaire (BIDQ): Assesses subjective dissatisfaction and interference caused by perceived appearance flaws.

Emotion Regulation Questionnaire (ERQ): Evaluates cognitive reappraisal and suppression strategies used to manage emotions.

Beck Depression Inventory-II (BDI-II): Measures depressive symptom severity.

Beck Anxiety Inventory (BAI): Measures general anxiety symptoms.

Data Analysis Plan ERP components will be analyzed using repeated-measures ANOVA, focusing on pre-post changes within and between groups. GSR data will be analyzed through paired and independent sample t-tests comparing skin conductance response and recovery. Eye-tracking data will be evaluated using linear mixed-effects models to identify patterns in fixation and gaze shifts.

Changes in psychometric scores will be analyzed via paired t-tests and ANCOVAs. Correlation analyses will examine the association between clinical improvement and physiological markers (e.g., reduced BDD-YBOCS scores and normalized alpha asymmetry). The statistical threshold will be set at p < .05, and all analyses will follow an intention-to-treat approach.

Scientific and Clinical Contribution This study represents a novel integration of CBT with multi-modal neurophysiological measurement in the context of BDD. It seeks to identify treatment-sensitive biomarkers of emotional and attentional regulation that may serve both diagnostic and therapeutic purposes. If successful, the findings will contribute to the development of personalized CBT interventions guided by real-time physiological feedback and objective clinical markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Body Dysmorphic Disorder (BDD) according to DSM-5 criteria
* Right-handed (to ensure consistency in EEG lateralization analyses)
* Minimum education level of high school (for questionnaire comprehension)
* Normal or corrected-to-normal vision (for eye-tracking calibration)
* Willingness to participate in all therapy and assessment sessions
* Signed written informed consent

Exclusion Criteria:

* Current use of psychotropic medication
* Current or past psychotherapy within the last 6 months
* Diagnosis of schizophrenia, bipolar disorder, or substance use disorder
* Neurological disorders (e.g., epilepsy, traumatic brain injury)
* Active suicidal ideation or recent suicide attempt (within past 12 months)
* Pregnancy (due to possible changes in physiological readings)
* Any uncorrected visual impairments or eye conditions preventing eye-tracking
* Presence of metal implants or devices incompatible with EEG recording

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in EEG Responses to Appearance-Related Stimuli | Baseline, Week 12 (Post-treatment)
  Electroencephalographic (EEG) responses to appearance-related stimuli will be analyzed as a composite neurophysiological outcome, integrating the following components:
  N170 (early facial processing), P300 (attention allocation), Late Positive Potential - LPP (emotional engagement), and Frontal Alpha Asymmetry (affective regulation). All EEG signals will be recorded using a 14-channel EEG system and processed through synchronized pipelines in iMotions, MATLAB, and R. Each ERP component will be extracted, cleaned, and averaged across trials. Although individual metrics will be analyzed separately for exploratory purposes, the primary analytic approach will treat these variables as a conceptually unified outcome representing neurophysiological change.
  Statistical comparisons will be conducted using repeated-measures MANOVA and linear mixed-effects modeling to evaluate the impact of CBT over time.
Change in Galvanic Skin Response (GSR) to Appearance-Related Stimuli | Baseline, Week 12 (Post-treatment)
  Sympathetic nervous system activity will be measured using Galvanic Skin Response (GSR) during exposure to appearance-related stimuli. The outcome consists of two integrated components:
  Skin Conductance Level (SCL): baseline tonic arousal Skin Conductance Response (SCR): phasic reactivity to stimuli Both components will be simultaneously recorded using the iMotions platform, preprocessed in MATLAB, and statistically analyzed using R. Though each parameter will be evaluated individually, the primary outcome represents a composite measure of autonomic arousal regulation.
  CBT is expected to result in decreased SCR amplitude and faster return to baseline SCL, reflecting improved stress regulation.
Change in Visual Attention Patterns During Facial Stimulus Exposure | Baseline, Week 12 (Post-treatment)
  Visual attention responses will be measured using eye-tracking during exposure to self-related and appearance-based stimuli. The outcome includes the following integrated metrics:
  Fixation Duration (ms) Fixation Count (number) Saccade Frequency (number per second) Pupil Dilation (mm) These metrics will be collected via a Gazepoint GP3 eye-tracker, synchronized through iMotions, and analyzed in R and MATLAB. While each measure will be analyzed individually in secondary analyses, this outcome collectively reflects attentional allocation and hypervigilance. CBT is expected to reduce biased attention toward self-perceived flaws and normalize gaze patterns.

SECONDARY OUTCOMES:
Change in BDD Symptom Severity: Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder / YBOCS-BDD | Baseline, Week 12
  The Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS) is a clinician-administered rating scale that assesses the severity of BDD-related obsessions and compulsions. It includes 12 items, each rated from 0 (no symptoms) to 4 (extreme symptoms), resulting in a total score range of 0 to 48. Higher scores indicate greater symptom severity.
Change in Body Image Disturbance Questionaire (BIDQ) | Baseline, Week 12
  he Body Image Disturbance Questionnaire (BIDQ) is a 7-item self-report questionnaire that assesses dissatisfaction with appearance, associated distress, and functional impairment. Each item is rated on a Likert scale from 1 to 5, with total scores ranging from 7 to 35. Higher scores reflect more severe body image disturbance.
Change in Emotion Regulation Questionaire (ERQ) | Baseline, Week 12
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report questionnaire measuring two emotion regulation strategies: cognitive reappraisal (6 items) and expressive suppression (4 items). Each item is rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Subscale scores range from 6 to 42 (reappraisal) and 4 to 28 (suppression). Higher scores reflect greater use of the respective strategy.
Change in Depressive Symptoms (Beck Depression Inventory-II) | Baseline, Week 12
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report questionnaire designed to assess the severity of depressive symptoms over the past two weeks. Each item is rated on a 4-point scale from 0 to 3, resulting in a total score range of 0 to 63.
  Higher scores indicate greater severity of depressive symptoms.
Change in Anxiety Symptoms (Beck Anxiety Inventory) | Baseline, Week 12
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionnaire designed to assess the severity of anxiety symptoms experienced during the past week. Each item is scored on a 4-point scale from 0 (not at all) to 3 (severely), yielding a total score range of 0 to 63.
  Higher scores reflect more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Selami Varol Ülker, Phd, Study Director — Üsküdar University; Gökben Hızlı Sayar, Prof, Study Chair — Üsküdar University; Eda Yılmazer, Phd, Principal Investigator — Beykoz University
Locations (1):
- Üsküdar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the primary and secondary outcomes of this trial (including EEG, GSR, eye-tracking data, and psychometric measures such as BDD-YBOCS, BIDQ, ERQ, BDI-II, and BAI) will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: Qualified researchers with a methodologically sound proposal and ethical approval may request access. Requests should be submitted to the corresponding author. Data will be shared through secure institutional platforms, and users must agree to terms of use that ensure participant confidentiality.